CLINICAL TRIAL: NCT03791632
Title: Oral Health Knowledge and Practice Among 8-9 Years Old Children.
Brief Title: Oral Health Among Children
Acronym: OHAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: RECHMPL18_0386
Record Dates: First submitted 2018-12-18; First posted 2019-01-02 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Schoolboy

STUDY DESIGN:
Intervention Model Description: 1. Test group
  2. Classes with a classical lecture style presentation
  3. classes with an intervention in the form of fun workshops on different themes by small groups of schoolchildren (8-10 children per workshop)
  4. classes with digital media intervention
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- witness (No Intervention): 2 control CE2 classes without oral sensitization actions
- group intervention 1 (Experimental): 2 CE2 classes with a classical lecture style presentation
  Interventions: Other: classical lecture style presentation
- group intervention 2 (Experimental): 2 CE2 classes with an intervention in the form of fun workshops on different themes by small groups of schoolchildren (8-10 children per workshop)
  Interventions: Other: an intervention in the form of fun workshops
- group intervention 3 (Experimental): 2 CE2 classes with digital media intervention
  Interventions: Other: digital media intervention

INTERVENTIONS:
Other: classical lecture style presentation — classical lecture style presentation
  Arms: group intervention 1
Other: an intervention in the form of fun workshops — an intervention in the form of fun workshops on different themes by small groups of schoolchildren (8-10 children per workshop)
  Arms: group intervention 2
Other: digital media intervention — digital media intervention
  Arms: group intervention 3

SUMMARY:
The aim of this study is to identify the knowledge and behavior on dental health and hygiene among adolescents. In most cases, the investigators know tooth decay can be prevented and reversed at an early stage by observing good oral hygiene. Few studies have been done among adolescents.

This study could justify the implementation of public health actions in terms of prevention.

ELIGIBILITY:
Inclusion criteria:

- All children of classrooms selectionned

Exclusion criteria:

- Children absent on the day of the intervention

Ages: 7 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 240 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
comparison of children's notes before and after a prevention intervention | 1 day
  The main result will be calculated with the total score to the questions. Each question corresponds to a point. The minimum score is 0 and the maximum score is 25.
  We will compare the evolution of the averages obtained by the control group and by all three other groups with Student test

OTHER OUTCOMES:
Compare the evolution of children's grades according to the type of intervention | before and after the explanation as well as one month and 6 months after the intervention
  For the secondary objective, we will compare the evolution of the averages obtained between the three groups with intervention with ANOVA test.
  Each question corresponds to a point. The minimum score is 0 and the maximum score is 25.
  before and after the explanation as well as one month and 6 months after the intervention
Determine the timeframe by which children forget the information they have been given | before and after the explanation as well as one month and 6 months after the intervention
  A questionnaire to know the oral knowledge will be distributed to the children before and after the explanation as well as one month and 6 months after the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Camille INQUIMBERT, PhD student, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC